CLINICAL TRIAL: NCT03431129
Title: Hyperpolarized 129Xe Magnetic Resonance Imaging for Evaluation of Radiation-Induced Lung Injury in Subjects Undergoing Thoracic Irradiation
Acronym: RILI
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment and not enough funding
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Giles Santyr, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000056200
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Radiation Induced Lung Injury (RILI)
Keywords: Xenon MRI, Lung, Radiation Induced Lung Injury,

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Hyperpolarized gas and proton lung MRI — Lung MRI for participants undergoing radiation therapy (RT)

SUMMARY:
The purpose of this work is to perform hyperpolarized (HP) 129Xe MRI in human subjects undergoing thoracic radiation therapy (RT), both before, during and following RT. HP 129Xe MR images will be analysed to provide maps of ventilation (V), perfusion (Q), apparent diffusion coefficient (ADC) and gas exchange. These results will be combined to yield a new measure of RILI, (i.e. dose volume histograms; DVHV/Q) and compared with conventional dose volume histograms (DVH), pulmonary function tests (PFTs), quality of life (QOL) questionnaire and CT measurements for assessment of RILI at each time point. The aim is to development a novel method for early and more sensitive method of detecting RILI before irreversible lung damage happens.

DETAILED DESCRIPTION:
Briefly, at the beginning of an approximate three hour study visit, the qualified investigator (QI) / delegate will explain the study procedure to the participants and the participants will have an opportunity to ask questions regarding the study procedure. Following the explanation of the study, written informed consent will be collected. During the study visit, participants will undergo: 1) brief medical history and clinical examination, 2) full pulmonary function tests, 3) proton MRI, 4) HP 129Xe MRI. Qualified research team members will perform a clinical examination on the participant to record their vital statistics like age, gender, height, weight, heart rate, respiratory rate, oral temperature and blood pressure. The QI/delegate, during a brief conversation with the participant, will collect relevant medical history from the participant to make sure the participant meets all the inclusion/exclusion criteria for the study. The QI will also make sure that the participant understands the study procedure and is willing to participate in the study. At each study visit at SickKids, the QI or delegate will also administer the QOL questionnaire to the participant. Based on the clinical examination results, medical history and the pulmonary function test results, the QI/delegate will determine if all the inclusion/exclusion criteria are met to proceed with the MRI part of the study visit.

ELIGIBILITY:
Inclusion Criteria:a) Patients 18 years of age or older; b) Diagnosis of locally advanced lung/esophageal/laryngeal or other type of cancer requiring radical intent RT to the thorax (with or without concurrent chemotherapy), consisting of 1.8 - 2 Gy daily fractions delivered over 5 - 6 weeks; c) Eastern Cooperative Oncology Group performance status 0 or 1; d) Preserved lung function as determined by a forced expiratory volume in 1 second (FEV1) > 70% to exclude patients with existing respiratory disorders (e.g. COPD, asthma etc.)

Exclusion Criteria:a) Planned anti-cancer surgery after radical RT; b) Chronic use of corticosteroids; c) Any previous RT to the thorax; d) History of ataxia telangiectasia or other known conditions that may increase radio-sensitivity; e) Planned for other anticancer therapy apart from RT or concurrent chemotherapy/RT f) Currently pregnant or lactating; g) Psychiatric or addictive disorders that would preclude obtaining informed consent or adherence to protocol; h) Inability to travel to obtain MRI scans; i) Any contraindications to MRI including but not limited to severe claustrophobia, implanted devices, aneurysm clips, neurostimulators (patients will be prescreened prior to registration).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant will be recruited from Princess Margaret Hospital, Toronto, Ontario and Juravinski Cancer Centre, Hamilton, Ontario.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
DVHV/Q | 2 years
  In-house software will be used to generate the ventilation, perfusion and gas exchange maps and calculate DVHV/Q

CONTACTS AND LOCATIONS:
Overall Officials: Giles Santyr, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared between the three participating sites in the study. A data transfer agreement has been implemented to enable this transfer smoothly.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after enrolling the first participant and will be available for the duration of the study